CLINICAL TRIAL: NCT04159376
Title: Assessment of the Accuracy of PET/MR in Detection and Monitoring Response of Bone Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0574-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Bone Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone Metastases Patients (Experimental)
  Interventions: Diagnostic Test: PET/MR

INTERVENTIONS:
Diagnostic Test: PET/MR — All patients will have a PET/CT and PET/MR study performed at the same clinical setting using a single dose of tracer administration.
  The study cohort includes 150 patients 18 years or older, having metastatic skeletal involvement on baseline PET/CT prior to treatment. Baseline studies and follow up studies of the patients referred post treatment, will be reviewed.
  The tracers will be FDG, labelled PSMA labelled Somatostatin and F-DOPA in order to assess skeletal lesions detection of all tumor types.
  Skeletal lesions will be divided into marrow-based lesions, lytic, blastic and scleroric lesions. Tracer uptake will be measured at baseline and after treatment. Metabolic PET parameters, CT appearance and MR parameters will be assessed.
  The best MR-based attenuation algorithm for detection of lesions and monitoring response will be derived.

SUMMARY:
The great promise of PET/MR for assessment of skeletal metastatic involvement is derived from the extensive experience with stand- alone MR, but initial data on the use of PET/MR for assessment of bone pathology indicate that PET/MR introduces unique issues that should be addressed when determining its role in this clinical scenario.

In this study cohort includes 150 patients 18 years or older, having metastatic skeletal involvement on baseline PET/CT prior to treatment. Baseline studies and follow up studies of the patients referred post treatment, will be reviewed.

The main goal of the study is to asses the accuracy of PET/MR in detection and monitoring response of bone metastases.

ELIGIBILITY:
Inclusion Criteria:

150 patients having metastatic skeletal involvement on baseline PET/CT prior to treatment

Exclusion Criteria:

1. Age <18.
2. Pregnant or breast feeding patients.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-12-25 (Estimated); Primary Completion 2020-02-25 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
The investigators will report about the number of patients who preformed PET/MR for assessment of skeletal involvement as well as activity after treatment, | 1 year
  and also preformed in routine PET/CT and to optimize the algorithm of MR-based attenuated PET images.

IPD SHARING:
Plan to Share IPD: Undecided